CLINICAL TRIAL: NCT03014271
Title: The Impact of Sources of Strength, a Primary Prevention Youth Suicide Program, on Sexual Violence Prevention Among Colorado High School Students
Brief Title: Primary Prevention Youth Suicide Trial in Colorado High Schools Prevention Among Colorado High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: University of Rochester (Other); Texas Tech University (Other); Colorado Department of Public Health and Environment (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB201702833; 2016-U-0436 (Other: IRB-02); 1U01CE002841-01 (NIH); GRANT12174446 (Other Grant/Funding Number: Centers for Disease Control)
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Suicide; Sexual Violence
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sources of Strength Suicide (SOS) (Experimental): Receive Sources of Strength Suicide (SOS) Prevention Program
  Interventions: Behavioral: Sources of Strength (SOS) Prevention Program
- SOS Waitlist Control (Active Comparator): Delayed implementation of Sources of Strength Suicide Prevention Program after 16 months.
  Interventions: Behavioral: Sources of Strength (SOS) Prevention Program

INTERVENTIONS:
Behavioral: Sources of Strength (SOS) Prevention Program — Sources of Strength is an evidence based program for youth suicide that trains student key leaders to strengthen social connectedness and healthy norms school-wide and is listed on the National Registry of Evidence Based Programs and Practices (NREPP).

SUMMARY:
Sources of Strength is an evidence based program for youth suicide that trains student key leaders to strengthen social connectedness and healthy norms school-wide and is listed on the National Registry of Evidence Based Programs and Practices (NREPP). This project will expand the existing evidence base by evaluating Sources of Strength for sexual violence outcomes in a randomized controlled trial (RCT) in twenty-four high schools.

DETAILED DESCRIPTION:
At present few programs systematically address broader social-ecological factors such as school-wide norms and youth-adult connectedness that research identifies as major drivers of sexual violence. To address this gap, this application proposes a large-scale RCT evaluation of Sources of Strength to evaluate for sexual violence perpetration outcomes. Sources of Strength is an evidence based program for youth suicide that trains student key leaders to strengthen social connectedness and healthy norms school-wide and is listed on the National Registry of Evidence Based Programs and Practices (NREPP). This project will expand the existing evidence base by evaluating Sources of Strength for sexual violence outcomes, which has never been done before. Twenty-four high schools will be recruited and stratified (rural or urban) and randomly assigned to one of two conditions: (a) immediate Sources of Strength intervention, (b) wait-list for Sources of Strength Implementation after 16 months.

ELIGIBILITY:
Inclusion Criteria:

* high school student in participating school, parents did not withdraw from study

Exclusion Criteria:

* none

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Change in sexual violence perpetration measured by method of survey | Baseline; Month 24
  Sexual violence perpetration will be measured by method of survey as part of the Sources of Strength suicide prevention program
Change in suicidal behaviors measured by method of survey | Baseline; Month 24
  Suicidal ideation and behaviors will be measured by method of survey as part of the Sources of Strength suicide prevention program

CONTACTS AND LOCATIONS:
Overall Officials: Tomei Kuehl, MPA, Study Director — Colorado Department of Public Health
Locations (1):
- Colorado Department of Public Health and Environment, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wyman PA, Cero IJ, Espelage DL, Reif T, Mintz S, LoMurray S, Nickodem K, Schmeelk-Cone KH, Delgado A. RCT of Sources of Strength Testing Impact on Suicide Attempts and Tests of Moderation by Sexual Violence Victimization and Perpetration. Am J Prev Med. 2025 Mar;68(3):465-474. doi: 10.1016/j.amepre.2024.11.008. Epub 2024 Nov 29. PMID 39617103